CLINICAL TRIAL: NCT04573686
Title: Prognostic Value of Serum Erythropoietin Level,Ferritin Level and Fibrinogen in Adult Low Risk MDS
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Asmaa Gamal Mohamed Abd Elaal, resident doctor, Assiut University
Other Study IDs: MDS
Record Dates: First submitted 2020-09-28; First posted 2020-10-05 (Actual); Last update posted 2020-10-05 (Actual); Status verified 2020-09

CONDITIONS: MDS
MeSH Terms: interventions — Erythropoietin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Erythropoietin — Erythropoietin will be given subcutenous to all patients

SUMMARY:
1. assessment of the penefit of erythropoietin administration in decreasing the frequency of blood transfusion in adult low risk MDS
2. assessement of the clinical significance of the relationship between hyperfibrinogenemia and the prognosis of patients with low risk MDS
3. assessement of the association between serum ferritin levels and patient _reported aspects and symptomes

DETAILED DESCRIPTION:
The myelodysplastic syndromes (MDSs) are clonal hematopoietic stem cell disorders characterized by progressive peripheral cytopenia due to ineffective hematopoiesis and a variable risk of transformation into acute myeloid leukemia (AML) .

Clinically, they can range from variable grade of cytopenia to forms not different from AML.

World Health Organization (WHO) MDS classifications from 2002:

included refractory anemia (RA), refractory anemia with ring sideroblasts (RARS), refractory cytopenia with multilineage dysplasia (RCMD), RCMD and ring sideroblasts (RCMDRS), refractory anemia with excess blasts (RAEB), and MDS associated with isolated del(5q) The most recent 2016 WHO MDS classifications are slightly different and include MDS with single lineage or multilineage dysplasia, MDS with ring sideroblasts and single or multilineage dysplasia, MDS with excess blasts, and MDS with isolated del(5q) .

A key first-line treatment option for many patients with symptomatic anemia associated with lower-risk MDS is erythropoiesis-stimulating agents (ESAs) (e.g., epoetin alpha ordarbepoetinalpha),whichmayalsobecombinedwithgranulocyte colony-stimulating factor (G-CSF At least, four mechanisms are recognized to underlie pancytopenia in myelodysplastic syndromes. Based on ferrokinetic studies two distinct mechanisms can be distinguished: (1) hypoproliferative suppressed erythropoiesis and (2) hypoproliferative/ineffective erythropoiesis,The predictive variables for ESAs response in MDS should be divided into biological and clinical variables. Biological variables include: endogenous erythropoietin levels < 500 U/L and marrow blasts < 10%, IPSS low INT-1, diagnosis of refractory anemia, and normal karyotype. On clinical plane, transfusion independence and short duration of disease are positive prognostic factors of response to ESAS .

sEPO levels have not only been correlated with response to ESAs. Various studies have also examined whether sEPO levels affect duration of response and overall survival among patients treated with ESAs. Other studies have examined whether sEPO levels can affect response to non-ESA treatments According to International Working Group criteria, erythroid response is considered an increase in hemoglobin level to at least 115 g/L without transfusion need. An increase in hemoglobin level of 15 g/L for patients with non-transfused anemia, or an abolished transfusion need, defines the criteria for partial response. To date, there is only a study assessing that Binocrit (Biosimilar epoetin alfa) is promising for the treatment of anemia of MDS patients. ER positively correlates with improvements in patients' cognitive status and positive changes in QOL after a median time of 2 years, 50% of patients may lose responsivenes to ESAs. Many factors, including depletion of iron, progression to acute myeloid leukemia, may be the underlying cause of loss responsiveness to ESAs. The first study evaluating the duration of response to erythropoietin in MDS patients Serum ferritin (SF) level represents a well-known indicator of the body's iron stores and inflammation. SF is commonly used as a marker of iron overload (defined as SF1000 ng/ mL) but this role has been often questioned, as SF value can be affected by acute infections, inflammations, and even malignant conditions, so that it is also considered as an acute phase protein. Several studies have evaluated tests other than the evaluation of SF level to estimate iron overload, such as Magnetic Resonance Imaging (MRI) and Superconducting Quantum Interference Device (SQUID) biomagnetic liver susceptometry Elevated SF levels represent a common condition among patients with myelodysplastic syndromes (MDS) and appears to be largely related to red blood cell (RBC) transfusion-dependence. However, iron overload is also present among many patients after MDS diagnosis and before RBC transfusion Fibrinogen is a protein produced following inflammation,and hyperfibrinogenemia is known as a poor prognostic factor in various tumors. In recent years, it has also been reported that hyperfibrinogenemia is a poor prognostic factor in diffuse large B-cell lymphoma.

However, whether hyperfibrinogenemia is a prognostic factor in patients with lower-risk myelodysplastic syndromes (MDS) remains unclear

ELIGIBILITY:
Inclusion Criteria:

* the participants are :adult low risk(IPSS score (2-3) myelodysplastic patients with median age (40-60)

Exclusion Criteria:

* patients with hiigh and intermediate risk MDS

Ages: 40 Years to 60 Years | Sex: All
Age Groups: Adult
Study Population: the participants are :adult low risk(IPSS score (2-3) myelodysplastic patients with median age (40-60)
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-01-01 (Estimated); Primary Completion 2022-01-01 (Estimated); Study Completion 2022-05-01 (Estimated)

PRIMARY OUTCOMES:
effect of erythropoietin on MDS prognosis | 1 year

REFERENCES:
- [Background] Gangat N, Patnaik MM, Tefferi A. Myelodysplastic syndromes: Contemporary review and how we treat. Am J Hematol. 2016 Jan;91(1):76-89. doi: 10.1002/ajh.24253. PMID 26769228
- [Background] Tefferi A, Vardiman JW. Myelodysplastic syndromes. N Engl J Med. 2009 Nov 5;361(19):1872-85. doi: 10.1056/NEJMra0902908. No abstract available. PMID 19890130
- [Background] Vardiman JW, Harris NL, Brunning RD. The World Health Organization (WHO) classification of the myeloid neoplasms. Blood. 2002 Oct 1;100(7):2292-302. doi: 10.1182/blood-2002-04-1199. PMID 12239137
- [Background] Cazzola M, Barosi G, Berzuini C, Dacco M, Orlandi E, Stefanelli M, Ascari E. Quantitative evaluation of erythropoietic activity in dysmyelopoietic syndromes. Br J Haematol. 1982 Jan;50(1):55-62. doi: 10.1111/j.1365-2141.1982.tb01890.x. PMID 6948570
- [Background] Della Porta MG, Malcovati L, Strupp C, Ambaglio I, Kuendgen A, Zipperer E, Travaglino E, Invernizzi R, Pascutto C, Lazzarino M, Germing U, Cazzola M. Risk stratification based on both disease status and extra-hematologic comorbidities in patients with myelodysplastic syndrome. Haematologica. 2011 Mar;96(3):441-9. doi: 10.3324/haematol.2010.033506. Epub 2010 Dec 6. PMID 21134982
- [Background] Stasi R, Abruzzese E, Lanzetta G, Terzoli E, Amadori S. Darbepoetin alfa for the treatment of anemic patients with low- and intermediate-1-risk myelodysplastic syndromes. Ann Oncol. 2005 Dec;16(12):1921-7. doi: 10.1093/annonc/mdi400. Epub 2005 Sep 15. PMID 16166176